CLINICAL TRIAL: NCT05504486
Title: A Phase 4, Multicenter, Single-arm, Open-label, Interventional fMRI Trial to Assess the Effect of Brexpiprazole as Adjunctive Therapy on Functional Brain Network Organization in Adults With Major Depressive Disorder and Symptoms of Anxiety
Brief Title: Open-label Brexpiprazole fMRI Trial in Adults With Major Depressive Disorder and Anxiety
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor strategic decision
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 331-201-00376
Record Dates: First submitted 2022-05-31; First posted 2022-08-17 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major depressive disorder (MDD); symptoms of anxiety; fMRI; brain networks; modularity; community structure; brexpiprazole; default mode network; salience network; central executive network; functional brain connectivity
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Brexpiprazole
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Oral tablet; take once daily; target daily dose of 2 mg

SUMMARY:
The purpose of this study is to use fMRI to evaluate the effects of brexpiprazole as add-on therapy to antidepressants on brain connectivity in individuals with MDD and symptoms of anxiety, aged 18 to 65.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 year of age
* Major Depressive Disorder (MDD) with symptoms of anxiety
* Stable treatment with less than 50% improvement

Exclusion Criteria:

* Contraindicated to perform fMRI scan
* Previous exposure to brexpiprazole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-29 (Estimated); Primary Completion 2023-03-22 (Estimated); Study Completion 2023-04-05 (Estimated)

PRIMARY OUTCOMES:
Change in fMRI resting-state salience network community structure from baseline to post-treatment | Week 6

SECONDARY OUTCOMES:
Association between change in resting-state salience network community structure and change in MADRS total score from baseline to post treatment. | Week 6
  Utilizing Jaccardized Czekanowski index
Change in Default Mode Network (DMN) community structure during emotional face viewing from baseline to post-treatment. | Week 6
  Utilizing Jaccardized Czekanowski index
Change in Central Executive Network (CEN) community structure during a working memory task from baseline to post-treatment. | Week 6
  Utilizing Jaccardized Czekanowski index

IPD SHARING:
Plan to Share IPD: No